CLINICAL TRIAL: NCT01638364
Title: Imaging Alcohol Induced Dopamine Release in the Human Brain: a PET/[11C](+)PHNO Study
Brief Title: Dopamine Release in the Human Brain Following Alcohol Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal Investigator; MD, PhD, CCFP, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 041/2012
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Heavy Drinking
MeSH Terms: interventions — Alcoholic Beverages; Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- alcoholic beverage (Active Comparator): 95% USP alcohol given at a dose of 1.5 g/l of body water mixed with orange juice and tonic water.
  Interventions: Drug: alcoholic beverage
- non-alcoholic beverage (Placebo Comparator): Orange juice and tonic water.
  Interventions: Drug: non-alcoholic beverage

INTERVENTIONS:
Drug: alcoholic beverage — An appropriate amount of 95% USP ethyl alcohol will be mixed in orange juice and tonic water to obtain a drink equivalent to 3-5 standard drinks. The beverage will be consumed over a period of 15 minutes.
  Other Names: Ethyl alcohol 95%
  Arms: alcoholic beverage
Drug: non-alcoholic beverage — This beverage will be a mixture of orange juice and tonic water. The beverage will be consumed over a period of 15 minutes.
  Other Names: Tropicana orange juice and Schweppes tonic water.
  Arms: non-alcoholic beverage

SUMMARY:
The purpose of this study is to examine whether there is an increase in dopamine levels in the human striatum following an oral administration of alcohol, as has been evidenced in animal models. This will be a Positron Emission Tomography (PET) study using the radiotracer, [11C]-(+)-PHNO (11C]-( + )-4-propyl- 3,4,4a,5,6,10b-hexahydro-2H-naphtho[1,2-b][1,4]oxazin-9-ol).

DETAILED DESCRIPTION:
This will be a within subjects study in 8 heavy drinkers ages 21-45. The within factors will be PET scans following an alcoholic beverage and following a non-alcoholic beverage. Participants will also have a baseline session prior to the scans where they will complete various cognitive tasks and questionnaires. During each PET scan, subjective drug effects as well as heart rate, blood pressure, blood alcohol content and cortisol levels will be collected. The change in PHNO binding potential between the two scan conditions will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of any ethnic origin between 21 and 45 years old.
* Reported consumption of at least two heavy drinking episodes (according to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) criterion of 5 drinks for males or 4 for females) in the past 30 days prior to assessment.
* Willing and capable to provide written informed consent
* Good command of the English language

Exclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis of alcohol dependence; receiving treatment for alcohol dependence
* Taking medications or have any medical condition for which alcohol is contraindicated
* Any medical condition requiring immediate investigation or treatment
* Previous head trauma/neurological condition such as clinically significant history of seizure disorder, a history of clinically significant head trauma (i.e., concussion resulting in clinically significant loss of consciousness) or past intracranial surgery
* Beck Depression Inventory score >16
* Current active or past suicidal ideation
* Pregnancy tested by urine and blood screen each PET study day or lactation
* Current DSM-IV diagnosis of any Axis I psychiatric disorder
* Regular use of any therapeutic or recreational psychoactive drug use during the last three months (with the exception of nicotine and alcohol) or other substance use disorder (including nicotine)
* Abnormal body mass (as defined as not within 20% of normal body mass index).
* Current past or anticipated exposure to radiation exceeding 20 mSv in the last year.
* Metal implants or paramagnetic objects within the body which may interfere with the magnetic resonance imaging (MRI).
* Claustrophobia or a history of panic attacks
* Abnormal clinical laboratory findings including serum creatinine greater than 2.0 mg/dl, abnormal liver function tests, elevated serum bilirubin (more than 1.5 times upper limit of normal), or pre-trial electrocardiogram (EKG) results demonstrating clinical significant abnormality

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in PHNO Binding Potential | 2 weeks
  Following the injection of the positron-emitting radiotracer [11C]-(+)-PHNO, binding of this radiotracer to dopamine receptors (DR) D2/3 will be measured using the PET scanner. As dopamine also binds to DR D2/3, either an increase or decrease in dopamine levels will either decrease or increase PHNO occupancy respectively. [11C]-(+)-PHNO binding potential will be measured on two different conditions (alcoholic beverage vs non-alcoholic beverage) on two separate days.

SECONDARY OUTCOMES:
Subjective effects of alcohol | 2 weeks
  During the PET scans, the subjective effects ( Alcohol Urges Scale, Biphasic Alcohol Effects Scale)of alcohol will be assessed at various time points throughout beverage consumption and PET scan.
Objective effects of alcohol | 2 weeks
  During the PET scans, the objective effects of alcohol (blood pressure, heart rate, blood alcohol content, blood cortisol levels) will be assessed at various time points throughout the drink consumption and PET scan.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Link Text: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research